CLINICAL TRIAL: NCT04489342
Title: An Investigation Into the Responsiveness of Inertial Measurement Unit (IMU) Sensor-based Tests in Measuring Changes in Spinal Mobility and Function in Axial Spondyloarthritis Patients Treated With Biologic Drug
Brief Title: Advanced Sensor Based Functional ASsessmenTs in Axial Spondyloarthritis
Acronym: ASFASTAS
Status: Recruiting | Type: Observational
Sponsor: Western Health and Social Care Trust (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, Dr Philip Gardiner, Consultant Rheumatologist, Western Health and Social Care Trust
Other Study IDs: WesternHSCT
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IMU sensor test — Measurement of maximum range of movement in the spine; Ambulatory observational data while performing standardised functional tests
  Other Names: ViMove (DorsaVi)

SUMMARY:
This is an observational study using Inertial Measurement Unit (IMU) sensors to measure the effects of biological therapy on spinal mobility and function in axial spondyloarthritis. Participants will undergo MRI scans before and after therapy in parallel to the sensor tests to establish correlation between changes in inflammatory signs and changes in spinal mobility.

DETAILED DESCRIPTION:
We will study 20 participants with active axial spondyloarthritis (axSpA) who are about to start biologic therapy as part of routine care. In brief, we will carry out the following assessments before and after therapy:

1. MRI of spine and Sacroiliac (SI) joints - modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) scoring
2. Record standard Patient recorded outcomes (PROs): Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Global (BASG), Bath Ankylosing Spondylitis Metrology Index (BASMI), Bath Ankylosing Spondylitis Functional Index (BASFI), Ankylosing Spondylitis Disease Activity Score (ASDAS), Ankylosing Spondylitis Disease Activity Score Health Index (ASAS-HI), Euroquol 3 level health assessment (EQ5D-3L), work productivity and activity impairment questionnaire (WPAI), Short QUestionnaire to ASsess Health enhancing physical activity (SQUASH),
3. Erythrocyte sedimentation rate (ESR), C-reactive protein (CRP)
4. IMU sensor tests in clinic for range of motion (ROM) in cervical, thoracic and lumbar spine.
5. IMU sensor tests at home for standardised function testing

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of axial spondyloarthritis fulfilling ASAS classification criteria.
2. Age ≥18 years old and <80 years.
3. Fulfilment of local criteria for biologic therapy for axSpA.
4. The subjects should be able to read, write, understand and complete study questionnaires.
5. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Safety contra-indication for biologic drug therapy.
2. Severely restricted hip movement (less than 20 degrees rotation in either hip).
3. History of previous clinical (symptomatic) vertebral fracture.
4. History of previous spinal surgery.
5. History of previous hip replacement surgery.
6. Major scoliosis deformity (in the opinion of the investigator).
7. Safety contra-indication for MRI assessment.
8. Previous biologic agent within 2 months.
9. Pregnant or breast-feeding women.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with active axSpA (BASDAI >4, Spinal Pain VAS >4)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Change in composite IMU sensor based metrology index (IMU-ASMI) | 4 months
  Change in AxSpA metrology index based on sensor tests of Range of Movement (i.e. spinal mobility). Scale 0-10, with 10 being severe loss of spinal mobility.

SECONDARY OUTCOMES:
Change in Bath Ankylosing Spondylitis Metrology Index (BASMI) | 4 months
  Change in traditional metrology index of spinal mobility. Scale 0-10, with 10 being severe loss of spinal mobility.
Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 4 months
  Change in axSpA disease activity. BASDAI scale 0-10, 10 representing high disease activity
Change in Assessment of Spondyloarthritis International Society Response Criteria (ASAS20) | 4 months
  Change in axSpA disease activity response - 20% improvement is regarded as minimum improvement in at least three of Patient global assessment, Pain assessment, BASFI and Inflammation (last two questions of BASDAI)
Change in modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) | 4 months
  Change in MRI score of inflammation. Range 0-72 the sum of scores for 24 vertebral edges in the lumbar and cervical regions, higher represents more spinal damage.
Change in Bath Ankylosing Spondylitis Functional Index (BASFI) | 4 months
  Change in traditional questionnaire function assessment 0-10 scale, 10 representing a high degree of functional impairment
Change in Sit to Stand Test Scores | 4 months
  Change in standardised function score. Time taken to complete 5 sit to stand actions from a seated position on a chair at standard height.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gardiner, MD, Principal Investigator — Western Health and Social Care Trust
Locations (1):
- Department of Rheumatology, Altnagelvin Hospital, Londonderry, N.Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Willing to share details of results and analyses with other researchers